CLINICAL TRIAL: NCT05145816
Title: A Dose-Finding and Proof-of-Concept Phase 1/2a Study of Belantamab Mafodotin in Relapsed or Refractory AL Amyloidosis
Brief Title: Phase 1/2a Study of Belantamab Mafodotin in Relapsed or Refractory AL Amyloidosis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Larry Anderson, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SCCC-06A21; STU-2021-0952
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: AL Amyloidosis; Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloidosis | interventions — belantamab mafodotin

STUDY DESIGN:
Intervention Model Description: This is an open-label, dose-escalation trial consisting of two parts: a Part 1 dose escalation phase and a Part 2 cohort expansion phase for safety and clinical activity testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort (DL 0) for Part 1 (Experimental): Cohort (DL 0) for Starting Dose : 1.9 mg/kg Belantamab mafodotin intravenously every 8 weeks
  Interventions: Drug: Belantamab mafodotin 1.9 mg/kg (8 weeks)
- Cohort (DL +1) for Part 1 (Experimental): Cohort (DL +1) for Dose Escalation: 2.5 mg/kg Belantamab mafodotin intravenously every 8 weeks
  Interventions: Drug: Belantamab mafodotin 2.5 mg/kg (8 weeks)
- Cohort (DL -1) for Part 1 (Experimental): Cohort (DL -1) for Dose De-escalation : 1.9 mg/kg Belantamab mafodotin intravenously every 12 weeks
  Interventions: Drug: Belantamab mafodotin 1.9 mg/kg (12 weeks)
- Cohort (DL -2) for Part 1 (Experimental): Cohort (DL -2) for Dose De-escalation: 1.4 mg/kg Belantamab mafodotin intravenously every 12 weeks
  Interventions: Drug: Belantamab mafodotin 1.4 mg/kg (12 weeks)
- Cohort Dose Expansion for Part 2 (Experimental): Cohort Dose expansion for Part 2: Belantamab mafodotin Dose from1.0 mg/kg to 2.5mg/kg every 4 weeks, 6 weeks, 8 weeks, or 12 weeks as determined by Part 1 recommended dosage calculations.
  Interventions: Drug: Belantamab mafodotin every 4 weeks, 6 weeks,8 weeks, or 12 weeks as determined by Part 1 recommended dosages
- Cohort (DL -3) for Part 1 (Experimental): Cohort (DL -3) for Dose De-escalation: 1.0 mg/kg Belantamab mafodotin intravenously every 12 weeks
  Interventions: Drug: Belantamab mafodotin 1.0 mg/kg (12 weeks)

INTERVENTIONS:
Drug: Belantamab mafodotin 2.5 mg/kg (8 weeks) — 2.5 mg/kg IV Belantamab mafodotin IV every 8 weeks for Part 1
  Arms: Cohort (DL +1) for Part 1
Drug: Belantamab mafodotin 1.9 mg/kg (8 weeks) — 1.9 mg/kg IV Belantamab mafodotin IV every 8weeks for Part 1
  Arms: Cohort (DL 0) for Part 1
Drug: Belantamab mafodotin 1.4 mg/kg (12 weeks) — 1.4 mg/kg Belantamab mafodotin IV every 12 weeks for Part 1
  Arms: Cohort (DL -2) for Part 1
Drug: Belantamab mafodotin 1.9 mg/kg (12 weeks) — 1.9 mg/kg Belantamab mafodotin IV every 12 weeks for Part 1
  Arms: Cohort (DL -1) for Part 1
Drug: Belantamab mafodotin every 4 weeks, 6 weeks,8 weeks, or 12 weeks as determined by Part 1 recommended dosages — Belantamab mafodotin Dose 1.0 mg/kg, 1.4 mg/kg, 1.9mg/kg or 2.5mg/kg every 4 weeks, 6 weeks, 8 weeks or 12 weeks as determined by Part 1 recommended dosages.
  Arms: Cohort Dose Expansion for Part 2
Drug: Belantamab mafodotin 1.0 mg/kg (12 weeks) — 1.0 mg/kg Belantamab mafodotin IV every 12 weeks for Part 1
  Arms: Cohort (DL -3) for Part 1

SUMMARY:
The goal of this study is to test the safety of drug, Belantamab Mafodotin, and see what effects (good and bad) it has on people who take it and amyloidosis, and to determine the most effective dose of the drug.

The study will have 2 phases (parts). The first phase of the study will test different doses of Belantamab Mafodotin. The second phase will test Belantamab Mafodotin at the dose level found to be safe and effective in phase 1

DETAILED DESCRIPTION:
Amyloid light chain amyloidosis (AL amyloidosis, ALA) is a rare plasma cell dyscrasia with an incidence ranging from 9.7-14.0 cases per million person-years. 75% of patients have cardiac involvement at diagnosis as evaluated by plasma cardiac biomarkers. The most common cause of morbidity and mortality is cardiac dysfunction.

Belantamab mafodotin has not been evaluated previously in patients with AL amyloidosis. Although Belantamab mafodotin has previously been or is currently being evaluated in patients with relapsed multiple myeloma (MM), these MM studies do not enroll participants with clinically significant cardiac dysfunction.

ALA represents a new patient population and therapeutic indication where patients invariably will have clinically significant cardiac, renal or other organ dysfunction at study enrollment. Therefore, the Phase I/IIa RRAL study will be comprised of two parts:

Part 1 - Dose Exploration (Escalation) this will be conducted to identify and select an appropriate dose of Belantamab mafodotin in regard to safety, as well as a preliminary evaluation of hematological and organ response. Part 1 will enroll a minimum of 3 to maximum of 18 patients, per dose cohort, and will be guided using the Bayesian optimal interval (BOIN) design.

Part 2 - Dose Cohort Expansion this will be an expansion cohort to further define the depth and durability of both hematological and organ response in 19 additional patients for a total of up to 37 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Participants medically diagnosed with relapsed or refractory Amyloid Light Chain Amyloidosis (AL amyloidosis) with one or more line of treatment as below:

   1. Must have received a proteosome inhibitor, alkylator and anti-cluster of differentiation 38 (CD38) antibody (e.g., daratumumab - for patients who were eligible to receive in newly diagnosed AL Amyloidosis) and autologous stem cell transplant (for transplant eligible candidates).

      OR
   2. Failed treatment and/or intolerant/ineligible for above agents

   NOTE: Patients who fail to achieve Partial Hematological Response or better after 2 cycles of induction therapy for newly diagnosed AL Amyloidosis are also eligible.
2. Participant must be over 18 years of age inclusive, at the time of signing the informed consent.
3. Participant and Disease Characteristics: Patient must have primary systemic AL amyloidosis, histologically confirmed at the initial diagnosis before initiation of 1st-line treatment by positive Congo red stain with green birefringence on polarized light microscopy, Or characteristic appearance by electron microscopy AND confirmatory AL amyloid typing (mass spectrometry-based proteomic analysis or immunofluorescence).
4. Patient must have measurable disease within 28 days prior to registration; serum quantitative immunoglobulins (immunoglobulin G (IgG), immunoglobulin A (IgA), and immunoglobulin M (IgM), serum free kappa and lambda, and serum protein electrophoresis (SPEP) with M-protein quantification must be obtained within 14 days prior to registration.
5. Measurable disease of amyloid light chain amyloidosis as defined by at least One of the following:

   1. Serum M-protein ≥0.5 g/dL by protein electrophoresis (routine serum protein electrophoresis and immunofixation).
   2. Serum free light chain ≥50 mg/L with an abnormal kappa: lambda ratio or the difference between the involved and uninvolved free light chains (dFLC) ≥50 mg/L.
6. One or more organs impacted by AL Amyloidosis according to consensus guidelines below per National Comprehensive Cancer Network (NCCN)Guidelines Version 1.2016:

   a. Cardiac Involvement i. Mean left ventricular wall thickness on echocardiogram greater than or equal to 12 mm in the absence of hypertension or valvular heart disease, OR N-terminal fragment brain natriuretic protein (NT-pro) brain natriuretic peptide (BNP) greater than 332 ng/mL provided that patient does not have impaired renal function (as defined by calculated creatinine clearance less than 25 mL/min) within 14 days prior to registration, OR prior cardiac biopsy (at time of diagnosis) showing amyloid deposition with past documented or presently noted clinical symptoms and signs supportive of a diagnosis of heart failure in the absence of an alternative explanation for heart failure.

   b. Non-Cardiac Organ Involvement

   i. Kidney: albuminuria greater than or equal to 500 mg per day on a 24-hour urine specimen within 35 days prior to registration, OR prior kidney biopsy (at the time of diagnosis) showing amyloid deposition.

   ii. Liver: hepatomegaly (total liver span > 15 cm) as demonstrated by computed tomography (CT) or magnetic resonance imaging (MRI) within 35 days prior to registration OR alkaline phosphatase (ALP) greater than 1.5 times the institutional upper limit of normal within 14 days prior to registration, OR prior liver biopsy (at the time of diagnosis) showing amyloid deposition.

   iii. Gastrointestinal tract: direct biopsy verification with symptoms.

   iv. Lung: biopsy verifications with symptoms and interstitial radiographic pattern.

   v. Soft tissue: tongue enlargement, clinical, arthropathy, claudication, presumed vascular amyloid, skin involvement, carpal tunnel syndrome, myopathy by biopsy or pseudohypertrophy.
7. Patients must have completed other systemic therapy or investigational drug > 28 days or five half-lives prior to registration, surgery (other than biopsies) > 28 days prior to registration, and any autologous stem cell transplant (ASCT) > 100 days prior to registration.
8. Patients must have a complete medical history and physical exam within 14 days prior to registration.
9. New York Heart Association (NYHA) Class 1 - 3a which has been clinically stable for 56 days before registration
10. Eastern Cooperative Oncology Group (ECOG) performance score 0, 1 or 2
11. Left ventricular ejection fraction (LVEF) by echocardiogram (ECHO) > 35% within 28 days prior to registration.
12. Adequate organ system functions within 14 days of registration as defined by the laboratory assessments below:

    a) Hematologic i) Absolute neutrophil count (ANC): ≥1.0 × 109/ L * ii) Hemoglobin: ≥8.0 g/dL * iii) Platelets: ≥50 × 109/L *

    b) Hepatic i) Total bilirubin: 1.5 × upper limit of normal (ULN); (Isolated bilirubin ≥1.5 × ULN is acceptable if bilirubin is fractionated, and direct bilirubin is <35%) ii) Alanine aminotransferase (ALT): ≤2.5 × ULN

    c) Renal i) Estimated glomerular rate (eGFRª): ≥30 mL/min/1.73 m2 Note: Laboratory results obtained during Screening should be used to determine eligibility criteria. In situations where laboratory results are outside the permitted range, the investigator may re-test the participant and the subsequent within range screening result may be used to confirm eligibility.

    * Without growth factor or cell transfusion support for the past 14 days prior to testing, excluding erythropoietin.

    ª As calculated by Modified Diet in Renal Disease (MDRD) formula (Appendix 4 in Protocol)
13. Females of childbearing potential: These participants must have a negative baseline pregnancy test within 72 hours prior to registration; this may be either a serum or urine pregnancy test, with a sensitivity of at least 50 milli-International unit (mIU)/mL; females of childbearing potential must also agree: (1) to have a pregnancy test prior to the start of each treatment cycle and (2) to either commit to continued abstinence from heterosexual intercourse or to use effective contraception while receiving study drug and for at least 4 months after receiving the last dose of study drug; females are considered to be of childbearing potential if they have had menses at any time in the preceding 24 consecutive months; in addition to routine contraceptive methods, effective contraception also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, she is responsible for beginning contraceptive measures.

    1. Is a woman of child bearing potential (WOCBP) and using a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency (as described in Appendix 9), during the intervention period and for at least 4 months after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.
    2. A WOCBP must have a negative serum pregnancy test (as required by local regulations) within 72 hours before the first dose of study intervention.
    3. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with a nearly undetected pregnancy.
    4. Non-childbearing potential is defined as follows (by other than medical reasons):

    i. ≥45 years of age and has not had menses for >1 year.

    ii. Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation.

    iii. Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.
14. Male participants are eligible to participate if they agree to the following during the intervention period and for 6 months after the last dose of study treatment to allow for clearance of any altered sperm:

    1. Refrain from donating sperm

       Plus, either:
    2. be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent

       Or
    3. agree to use a barrier method of birth control (e.g., male condom), even if they have undergone a successful vasectomy, and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year as when having sexual intercourse with a woman of childbearing potential (including pregnant females).
15. Patients with Human Immunodeficiency Virus (HIV) infection are eligible if:

    1. patients without a history of Acquired Immune Deficiency Syndrome (AIDS)-defining opportunistic infections
    2. patients with a history of AIDS-defining opportunistic infection may be eligible if they have not had an opportunistic infection within past 12 months.
    3. Patients on active anti-retroviral therapy are eligible as long as anti-retroviral therapy is established for at least four weeks and have HIV viral load less than 400 copies/ml prior to enrollment.
16. Patients with chronic Hepatitis B Virus (HBV) infection or chronic Hepatitis C Virus (HCV) infection or virologically suppressed on HCV treatment are eligible if:

    1. Hepatitis B surface antigen (HBsAg)-negative, anti-Hemoglobin C (HBc)-positive patients are at lower risk of HBV reactivation compared with HBsAg-positive patients, risk of HBV reactivation should be considered in all patients and if patients can be on anti-HBV prophylaxis prior to initiation of anti-cancer therapy.
    2. Patients with chronic HBV infection with active disease who meet the criteria for anti HBV therapy should be on a suppressive antiviral therapy prior to initiation of cancer therapy.
    3. Patients actively on treatment for HCV should have HCV below the limit of quantification before initiation of anti-cancer therapy.
    4. Patients who are HCV antibody (Ab) positive but HCV Ribonucleic Acid (RNA) negative due to prior treatment or natural resolution of infection are eligible.

Exclusion Criteria:

1. Patients previously treated for active symptomatic multiple myeloma.
2. Any corneal disease except for mild epithelial punctate keratopathy.
3. Patients with known immediate or delayed hypersensitivity reaction or idiosyncratic reactions to belantamab mafodotin or drugs chemically related to belantamab mafodotin, or any of the components of the study treatment.
4. Patients eligible for autologous stem cell transplantation (ASCT).
5. Evidence of significant cardiovascular condition as specified below:

   1. N-terminal-prohormone of brain natriuretic peptide (NT-proBNP) ≥ 8500ng/L within 14 days of registration.
   2. New York Heart Association (NYHA) classification IIIB (3b) through IV (4) heart failure
   3. Heart failure that in the opinion of the investigator is on the basis of ischemic heart disease (e.g., prior myocardial infarction with documented history of cardiac enzyme elevation and electrocardiogram (ECG) changes) or uncorrected valvular disease and not primarily due to AL amyloid cardiomyopathy
   4. Unstable heart failure defined as emergency hospitalization for worsening, or decompensated heart failure, or syncopal episode within 1 month of screening
   5. Subjects with a history of sustained ventricular tachycardia or aborted ventricular fibrillation or with a history of atrioventricular nodal or sinoatrial (SA) nodal dysfunction for which a pacemaker/implantable cardioverter-defibrillator (ICD) is indicated but not placed (Subjects who do have a pacemaker/ICD are allowed on study)
   6. Interval from the Q wave on the ECG to point T using Fredericia's formula (QTcF) > 500 msec. Subjects who have a pacemaker may be included regardless of calculated QTc interval
   7. Symptomatic, clinically significant autonomic neuropathy which the Investigator feels will preclude administration of study treatment
   8. Acute coronary syndrome, or any form of coronary revascularization procedure including coronary artery bypass grafting (CABG), within 6 months of screening
   9. Prior solid organ transplant, or anticipated to undergo solid organ transplantation, or requiring left ventricular assist device (LVAD) implantation, during the course of the study
   10. Stroke within 6 months of screening, or transient ischemic attack (TIA) within 3 months of screening
   11. Evidence of current clinically significant uncontrolled arrhythmias, including clinically significant ECG abnormalities such as 2nd degree (Mobitz Type II) or 3rd degree atrioventricular (AV) block
   12. History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within three (3) months of Screening
   13. Uncontrolled hypertension
6. Prior history of malignancy with the exception of the following: adequately treated basal cell or squamous cell skin cancer, curatively treated non-melanoma skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for at least two years.
7. Presence of any comorbid or uncontrolled medical condition (e.g., diabetes mellitus or uncontrolled hypertension) at screening, which in the opinion of the investigator would increase the potential risk to the subject.
8. Unwillingness or inability to follow the procedures outlined in the protocol.
9. Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 4 weeks or five half-lives, whichever is shorter, before Cycle 1 Day 1.
10. Participant must not use contact lenses while participating in this study.
11. Participant must not have had major surgery ≤ 4 weeks prior to initiating study treatment.
12. Participant must not have any evidence of active mucosal or internal bleeding.
13. Participant must not have any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions (including lab abnormalities) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures.
14. Participants must not be pregnant or lactating.
15. Participant must not be simultaneously enrolled in any interventional clinical trial.
16. Participant must not have an active infection requiring treatment.
17. Participant must not have current unstable liver or biliary disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if otherwise meets entry criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety/Tolerability as measured by number of subjects with dose limiting toxicity (Part 1) | Up to 90 days after completing therapy
  Safety/Tolerability is measured by the number of participants treated with different dose level of belantamab mafodotin who experience dose limiting toxicity adverse events (AE) >= Grade 3, as defined by Common Terminology Criteria for Adverse Events by CTCAE v5.0 for Part 1.
Safety/Tolerability at the recommended Phase II dose of Belantamab Mafodotin, as measured by number of subjects with dose limiting toxicity (Part 2) | Up to 90 days after completing therapy
  Safety/Tolerability at the recommended Phase II dose of Belantamab Mafodotin is measured by the number of subjects who experience dose limiting toxicities (>= Grade 3, as defined by Common Terminology Criteria for Adverse Events by CTCAE v5.0) and cardiac and ocular AEs.

SECONDARY OUTCOMES:
Percentage of subjects with preliminary hematological responses associated with Belantamab mafodotin (Part 2) | Up to 2 years after the last dose
  Hematologic responses are assessed as the Overall Response Rate (ORR) which is the percentage of subjects with a confirmed partial response (PR) or better i.e. very good partial response (VGPR), complete hematological response (CHR). The criteria for : i) PR is - Baseline dFLC (difference between iFLC and uninvolved FLC) ≥ 50mg/L: A greater than 50% reduction in the dFLC, Baseline dFLC < 50 mg/L: ≥ 50% reduction in serum M-protein plus reduction in 24-hr urine M-protein by ≥ 90% or to <200 mg/24 hours ; ii) Very good partial response is - Baseline dFLC ≥ 50mg/L:Reduction in the dFLC<40mg/L, Baseline dFLC < 50 mg/L: ≥ 90% reduction in serum M-protein plus urine M-protein <100 mg/24 hours ; iii) CHR is - the normalization of free light chain (FLC) levels and ratio, negative serum and urine immunofixation (IFE)
Percentage of subjects with cardiac response associated with Belantamab mafodotin (Phase 2) | Up to 2 years after the last dose
  Cardiac Response is assessed as Overall Cardiac Response Rate (OcRR) which is the percentage of participants with a confirmed plasma NT-proBNP reduction from baseline of ≥ 30% .
Percentage of subjects with non-cardiac organ response associated with Belantamab mafodotin (Phase 2) | Up to 2 years after the last dose
  Non-Cardiac Organ Response (i.e. kidney and/or liver) assessed as: Organ response rate (OrRR) as defined as:
  1. Kidney: reduction in proteinuria by ≥ 30% from baseline; or, a reduction in proteinuria < 0.5g/24 hours without renal progression
  2. Liver: 50% decrease in abnormal alkaline phosphatase (ALP) from baseline
Percentage of participants with Complete Hematological Response (CHR) (Phase 2) | Up to 2 years after the last dose
  Complete Hematological Response (CHR), defined as normalization of the free light chain levels and ratio, negative serum and urine immunofixation
Duration of Response (DoR) (Phase 2) | From time of documented evidence of PR or better until PD or death due to PD in participants with confirmed PR or better, assessed up to 2 years after the last dose
  Duration of Response (DoR), defined as the time from first documented evidence of PR or better until progressive disease (PD) or death due to PD among participants who achieve confirmed PR or better. Progressive disease is defined using this criteria.
Time to Response (TTR) (Phase 2) | From time of start of therapy to the first documented evidence of response (PR or better), assessed up to 2 years after the last dose
  Time to Response (TTR), defined as the time between the start of therapy and the first documented evidence of response (PR or better) among participants who achieve confirmed PR or better.
Time to Best Response (TTBR) (Phase 2) | From time of earliest date of best response with confirmed PR or better, assessed up to 2 years after the last dose
  Time to Best Response (TTBR), defined as the time between the earliest date of achieving best response among participants with a confirmed PR or better.
Time to Progression (TTP) (Phase 2) | From time of start of therapy to the earliest date of documented hematological progression or death due to hematological progression, up to 2 years after the last dose
  Time to Progression (TTP), defined as the time from the start of therapy until the earliest date of documented hematological progression, or death due to hematologic progression, where hematologic progression is defined as one of the following: From complete hematological response (CHR), abnormal free light chain ratio (light chain ratio must double) or from CHR/VGPR/PR, 50% increase in serum M-protein to >0.5 g/dL or 50% increase in urine M-protein to >200 mg/day (a visible peak must be present) ; Involved Free light chain (iFLC) increase of 50% to >100 mg/L
Duration of Cardiac Response (DocR) (Phase 2) | From time of first documented evidence of a 30% reduction, or better, in plasma NT-proBNP until cardiac progression, up to 2 years after the last dose
  Duration of Cardiac Response (DocR), defined as the time from first documented evidence of a 30% reduction, or better, in plasma NT-proBNP until cardiac progression as defined as a > 30% & > 300 ng/L increase in plasma NT-proBNP; Or, > 75% increase in high-sensitivity (hs) cardiac troponin-T (cTnT).
Time to Cardiac Response (TTcR) (Phase 2) | From date of starting treatment and the first documented evidence of plasma NT-proBNP cardiac response, up to 2 years after the last dose
  Time to Cardiac Response (TTcR), defined as the time between the date of starting treatment and the first documented evidence of plasma NT-proBNP cardiac response.
Time to Cardiac Progression (TTcP) (Phase 2) | From date of starting treatment until the earliest date of documented cardiac disease progression or death due to progressive cardiac disease, up to 2 years after the last dose
  Time to Cardiac Progression (TTcP), defined as the time from the date of starting treatment until the earliest date of documented cardiac disease progression as defined above, or death due to progressive cardiac disease.

CONTACTS AND LOCATIONS:
Overall Officials: Larry Anderson, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (5):
- United States (5):
  - Stanford Cancer Institute, Stanford, California
  - Tufts Medical Center, Inc., Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No